CLINICAL TRIAL: NCT06266962
Title: Comparing the Efficiency of Two Prophylactic Approaches in Patients at Risk of Developing Intraoperative Floppy Iris Syndrome
Brief Title: Comparing the Efficiency of Two Approaches in Patients at Risk of Developing Intraoperative Floppy Iris Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Olomouc (Other)
Collaborators: Palacky University (Other)
Responsible Party: Principal Investigator, Zuzana Schreiberova, Principal Investigator, University Hospital Olomouc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3/24
Record Dates: First submitted 2024-02-07; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Intraoperative Floppy Iris Syndrome; Cataract; Age-related Cataract; Adrenergic Receptor Antagonist Adverse Reaction
Keywords: Intraoperative Floppy Iris Syndrome; Cataract; Age-related Cataract; Atropine; Epinephrine; Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Alpha1-adrenergic receptor antagonists; Tamsulosin
MeSH Terms: conditions — Cataract; Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Epinephrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1% Atropine drops (Active Comparator)
  Interventions: Drug: 1% Atropine drops
- Epinephrine (Active Comparator)
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: 1% Atropine drops — Patients administered 1% Atropine drops twice a day for a week before the cataract surgery.
  Arms: 1% Atropine drops
Drug: Epinephrine — Patients underwent the instillation of epinephrine into the anterior chamber at the beginning of the cataract surgery.
  Arms: Epinephrine

SUMMARY:
Intraoperative Floppy Iris Syndrome (IFIS) is a potentially serious cataract surgery complication. IFIS is most commonly associated with the chronic use of tamsulosin and other alpha1-adrenergic receptor antagonists prescribed in low urinary tract symptoms. There are a number of guidelines for operative technique modifications with the aim to prevent the development of IFIS. The study focuses on two options for prophylactic strategies: the application of atropine drops and the instillation of intracameral epinephrine.

DETAILED DESCRIPTION:
Intraoperative Floppy Iris Syndrome (IFIS) is a complication that may develop during cataract surgery. IFIS is most commonly associated with the chronic use of tamsulosin and other alpha1-adrenergic receptor antagonists prescribed in low urinary tract symptoms. It is characterised by an unstable iris whose increased elasticity may lead to a number of complications during cataract extraction with a negative impact on vision outcomes. Basic features of IFIS are a 'floppy' iris that 'ripples' in irrigation, insufficiently inducible mydriasis with progressive intraoperative miosis (despite repeated application of mydriatics) and the tendency of the iris to prolapse into the phacoemulsification probe.

IFIS is a complication that makes surgery more difficult for the eye surgeon. There is a risk of intraoperative conditions such as rupture of the posterior capsule with lens masses luxation into the vitreous body, damage to the iris by surgical instruments, damage to the endothelium with washout of endothelial cells, hyphaema, or prolapse of the vitreous body into the anterior chamber.

There are several surgical approaches to prevent the development of IFIS and facilitate easier management of the entire cataract extraction in unstable iris. The investigators recommend patients apply 1% atropine drops twice a day for one week during the pre-operative period. A more elegant method is the administration of epinephrine into the anterior chamber at the beginning of the cataract surgery. The aim of this study is to evaluate the effectiveness of two mydriatic agents - the administration of atropine drops and the instillation of epinephrine into the anterior chamber and to compare their effectiveness in preventing IFIS.

ELIGIBILITY:
Inclusion Criteria:

* age-related cataract
* age over 18 years
* men with diagnosed benign prostatic hyperplasia
* history of having taken, or currently taking any systemic α1-adrenergic receptor antagonists for low urinary tract symptoms
* performing of pre-operative examination before cataract surgery
* signed informed consent

Exclusion Criteria:

* presence of any pupil deformity due to e.g. post-traumatic condition
* iris defect of any aetiology
* status post anterior uveitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Development of IFIS | intraoperative
  Development of IFIS - yes/no.
Severity of IFIS | intraoperative
  Determination of severity of IFIS - mild/moderate/severe.
Incidence of intraoperative complications | intraoperative
  To find out if there are any intraoperative complications in either group (%) and what the complications are (rupture of the posterior capsule of the lens, intraoperative hypotonia, iris defect atc.)

CONTACTS AND LOCATIONS:
Overall Officials: Miroslava Maluskova, MD, FEBO, Principal Investigator — University Hospital Olomouc and Palacky University Olomouc
Locations (1):
- Department of Ophthalmology, University Hospital Olomouc, Olomouc, Czechia

REFERENCES:
- [Derived] Maluskova M, Maresova K, Schreiberova Z, Paskova B, Karhanova M. Comparing the efficiency of two prophylactic approaches in patients at risk of developing Intraoperative Floppy Iris Syndrome. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2025 Sep 19. doi: 10.5507/bp.2025.025. Online ahead of print. PMID 40977319